CLINICAL TRIAL: NCT05330104
Title: SENSE Study: Feasibility of Using Continuous, Remote Symptom Monitoring to Identify and Respond to Early Fall-risk for Patients With Chemotherapy-induced Peripheral Neuropathy
Brief Title: SENSE Study: Remote Symptom Monitoring for Patients With Chemotherapy-induced Peripheral Neuropathy
Acronym: SENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1830048-2
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mEMA Arm (Experimental): In this arm, participants will be using a mobile survey system to track the emergence of Chemotherapy-Induced Peripheral Neuropathy symptoms and fall risk over the course of the participant's chemotherapy.
  Interventions: Behavioral: Mobile Ecological Momentary Assessment

INTERVENTIONS:
Behavioral: Mobile Ecological Momentary Assessment — mEMA is a tool that allows for scheduled or triggered surveys to assess a participant's CIPN symptoms and/or fall risk
  Other Names: mEMA

SUMMARY:
The main purpose of this study is to determine the threshold level of lower extremity CIPN symptoms that put patients who have been prescribed a neurotoxic chemotherapy agent (e.g., paclitaxel, docetaxel, oxaliplatin or cisplatin) as part of their treatment regimen for cancer at-risk for falling. The investigators believe that by specifying early CIPN symptoms that predict fall-risk, The investigators will ultimately be able to identify at-risk patients who could be referred to rehabilitative services to prevent injurious falls while enabling them to continue the chemotherapy treatment that could save their lives.

DETAILED DESCRIPTION:
Patients who are treated with neurotoxic chemotherapy as part of their cancer treatment regimen often experience lower extremity chemotherapy-induced peripheral neuropathy (CIPN) that causes motor and sensory loss, which increases their fall risk. CIPN is a potential side-effect of many chemotherapy regimens used to treat the most common adult cancers. In fact, CIPN occurs in as many as 90% of cancer patients whose chemotherapy includes taxanes, vinca alkaloids, or platinum agents. The symptoms of CIPN affect balance, which may put patients at-risk for falls. While much of the research in this area pertains to participants with long-standing CIPN symptoms, most authorities explicitly advocate for early monitoring for symptoms of CIPN and for earlier intervention than is currently the standard of care. However, there is little scientific literature that specifies (1) when in patients' chemotherapy regimens these symptoms typically first reach a significant CIPN or fall/near fall symptom threshold, and (2) how to best systematically track symptom emergence. Further, there are no evidence-informed best practices for early identification of CIPN symptoms and grading of severity, nor is there clear information about early time-points for symptom emergence that could inform when clinicians should begin to pay attention to patients' fall risk.

To address this, a team of expert clinicians and researchers from Courage Kenny Rehabilitation Institute (CKRI) and Allina Health Cancer Institute (AHCI) will use a mobile survey system to track the emergence of CIPN symptoms and fall risk over the course of patients' chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 45 years old
2. New cancer diagnosis other than a primary brain tumor
3. A taxane and/or platinum chemotherapy agent has been prescribed as part of the treatment regimen for cancer.
4. English speaking
5. Able to see, hear, speak (with or without assistive devices)
6. Able to walk without an assistive device - for example: cane, walker, walking stick(s) at the start of cancer treatment
7. Able to provide own transportation to study visits
8. Willing and able to commit to symptom tracking three times weekly via mEMA for up to 9 months.
9. Owns a smartphone with one of the following operating system versions:

   iOS 8.0 - 8.4, 9.0 - 9.3, 10.0 - 10.3, 12, 13.3 or later Android 7.0 - 7.1.2, 8.0 - 8.1.0, 9, 10 or later
10. Agree to use personal smartphone to download the mEMA application and respond to application notifications.

Exclusion Criteria:

1. Individuals who started their chemotherapy regimen greater than 4 weeks prior to study enrollment.
2. Individuals being treated for a primary brain tumor

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with mEMA | Through study completion, up to 6 months
  Administer a mEMA Experience Survey at each in-person fall-risk assessment to obtain information about participant experience with mEMA over the course of the study.
Patient Adherence to mEMA | Through study completion, up to 6 months
  Conduct descriptive analyses (mean, mode, median) to determine adherence rates and patterns for mEMA adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gilchrist, PhD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No